CLINICAL TRIAL: NCT01089478
Title: Cells in the Lumbar Epidural Space of Patients With Low Back Pain and/or Radiculopathy
Brief Title: Cytology Study of Cells From Patients With Low Back Pain
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator passed away.
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Other Study IDs: L05-099
Record Dates: First submitted 2010-03-17; First posted 2010-03-18 (Estimated); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Back Pain
Keywords: Back pain; Low back pain; Cytology; Epiduroscopy; Pain; Radiculopathy
MeSH Terms: conditions — Back Pain; Low Back Pain; Pain; Radiculopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — During epiduroscopy up to five (5) specimen samples will be collected from different sites in the epidural space
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators are doing this study to learn more about the cause of back pain with or without pain shooting down one or both legs. The investigators specifically want to know if cells that move into injured areas of the body are present in a space in the spine (epidural space) of patients with back pain and with or without shooting pain. The investigators will collect cells when patients are being treated, then examine the cells using a microscope. The investigators also will shine different colors of light into the epidural space to see if there is a correlation between how different colors of light are reflected and the types of cells present.

DETAILED DESCRIPTION:
The objective of this study is to examine the cell population in the epidural space of patients with low back pain +/- radiculopathy to determine if the cell population reveals pathological processes sustaining the pain. Cells will be collected for microscopic inspection and will be examined in situ during exposure to white and UV light. The overall goal is to advance our knowledge about the etiology of low back pain +/- radiculopathy to guide mechanistic based therapy.

The primary information sought is to determine if description of pathological processes based upon direct observation with percutaneously placed epiduroscopes can be confirmed by cytological analysis. the observations described include: 1) increased fibrosis from slight to complete replacement of other tissue, or obliteration of the epidural space; 2) alteration of color and/or appearance of epidural fat; 3) increased or decreased vascularity. The overall description range from acute inflammatory changes to advanced fibrosis (scarring).

Specimens for cytological analysis will be obtained from different sites in the epidural space by using commercially available cytology specimen collecting brushes and/or catheters. These are inserted through the working channel of an epiduroscope into the lumbar epidural space to aid treatment.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form
* Age >18 years at the time of signing the informed consent form
* A diagnosis of low back pain with or without radiculopathy and scheduled for epiduroscopy assisted epidural neurolysis

Exclusion Criteria:

* Patients not scheduled for epiduroscopy assisted epidural neurolysis
* Are female who is pregnant
* Are a female of childbearing age and are not using an acceptable form of contraception
* Have a medical history or condition that would not make the patient a good candidate for epiduroscopy procedure
* Are unwilling or unable to provide written informed consent and/or to obey the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: consecutive patients receiving epidural neurolysis treatment for back pain
Sampling Method: Probability Sample
Enrollment: 605 (Actual)
Dates: Start 2005-04 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Characteristics of cell samples | 5 years
  The investigators expect that cell types identified will vary some from patient to patient depending in part upon how acute or chronic is the patient's disease and whether or not the patient has had prior surgery. The investigators expect the cells will indicate that a pathological process is present and will provide information about the characteristics of the process

SECONDARY OUTCOMES:
Reflect light | 10 years
  The investigators expect that different tissue types in the epidural space will reflect white light differently and that some cells involved in pathological processes will autofluoresce

CONTACTS AND LOCATIONS:
Overall Officials: James E Heavner, DVM, PhD, Principal Investigator — Texas Tech University Health Sciences Center